CLINICAL TRIAL: NCT01244841
Title: The Effect on 30 Day Health Status After Early Discharge in Patient With ST Elevation Myocardial Infarction Treated With Primary PCI
Brief Title: Effects on Health Status in Patients Early Discharged After Primary Percutaneous Coronary Intervention (PCI)
Acronym: INUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/807-4
Record Dates: First submitted 2010-10-12; First posted 2010-11-19 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Acute Myocardial Infarction
Keywords: ST elevation acute myocardial infarction; Primary percutaneous coronary intervention; Discharge; Health status; Quality of care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): Randomised to standard post MI care and length of hospital stay decided by treating physician.
- Early discharge (Active Comparator): Randomised patient where all post MI investigations, treatment, follow-up plans and information will be performed within 3 days, and the patients are thereafter discharged.
  Interventions: Procedure: fast post MI care

INTERVENTIONS:
Procedure: fast post MI care — All post MI investigations, treatment, start of medication, information are performed within 3 days after admittance.
  Arms: Early discharge

SUMMARY:
In patients with ST elevation myocardial infarction (STEMI)treated with primary percutaneous coronary intervention (PPCI) a subset with low risk for late complications can be identified. Early discharge (<72h) of these patients can compromise initiation of prophylaxis, information and other investigations. The researchers want to investigate prospectively whether early discharge compared to regular care have comparable patient centered outcomes at 30 days follow-up.

DETAILED DESCRIPTION:
The safety and feasibility of early discharge of low-risk STEMI treated with thrombolysis or PPCI patients have previously been investigated. It is possible to identify a subset of patients with very low risk for subsequent cardiac events in the short-term, where prolonged hospital stay beyond three days does not alter the outcome. Early discharge have however, not been included in STEMI management guidelines formally. The effects of this discharge regimen on STEMI patients' health status (symptoms, functional capacity and quality of life) is not previously investigated. Shorter hospital stays saves health care resources. On the other hand, short in-hospital stay can affect the perceived satisfaction of care. Initiation of medical treatment, patient education, life style counselling and follow-up routines may suffer. Additionally, early discharge can increase anxiety and symptom level reducing the health related quality of life (HRQOL) and also lead to readmission. Patient satisfaction has become a recognised measure of the quality of health care.Currently there is little information on how early discharge influence the patients' satisfaction with the health care or the subjective perceived of HRQOL after discharge. We therefore wish to perform a prospective trial comparing outcomes with regard to satisfaction of care and HRQOL in patients admitted for STEMI randomised to either early discharge or standard care.

ELIGIBILITY:
Inclusion Criteria:

* ST elevation acute myocardial infarction
* Undergoing primary PCI

Exclusion Criteria:

* Zwolle low risk criteria score >4
* Re-infarction, post AMI ischemia.
* Need for urgent repeat invasive procedures.
* Non-cardiac complication (bleeding, stroke oa.) or concomitant diseases likely to increase length of hospital stay.
* Patient or caring physician refuse to early discharge or study inclusion.
* Early discharge impossible due to social, nursing or family reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Evaluate whether the health status after early discharge compared to standard care is comparable in low-risk primary PCI patients. | 1 month
  This is an equivalence study comparing health related quality of life(HRQOL) and quality-of-care satisfaction between the 3 days stay and standard regimen groups at 30 days after AMI. The scores of the SF-36, Seattle Angina Questionaire and Hospital Anxiety & Depression Scale for patients in both study groups will be compared. The forms will be filled out by the patients at baseline and at 30 days follow-up.

SECONDARY OUTCOMES:
Comparison between the study groups of readmission rates within 1 month. | 30 days
Comparison between the study groups of compliance with, and target dosing of medical therapy. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Tor Melberg, MD PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Rogaland, Norway